CLINICAL TRIAL: NCT01158196
Title: Effect of Infra-red Diode Laser on Improvement of Surgical Scar and on the Prevention of Excised Keloids Recurrence-Pilot Study
Brief Title: Safety and Efficacy of Infrared Diode Laser on Improvement of Scar and Prevention of Recurrence of Excised Keloid
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ekkyo (Industry)
Responsible Party: Pr. Magalon/ Plastic Surgeon, APHM
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: E-200-M/keloid project; 2010-A00323-36 (Other: AFSSAPS - RCB ID NUMBER)
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Keloid; Surgical Scar
Keywords: laser; keloid; scar
MeSH Terms: conditions — Keloid; Cicatrix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- infra-red diode laser (Experimental): one session, one dose
  Interventions: Device: infra-red diode laser

INTERVENTIONS:
Device: infra-red diode laser — laser treatment of scar after keloid excision
  laser treatment of surgery scar

SUMMARY:
A pilot study will be conducted on 2 type of subjects, one with plastic surgery scar with a randomization of laser treated portions, and other with keloid excision scar with a complete laser treatment. The aim is to evaluate the infra-red diode laser influence on keloid recurrence and scar prevention. The keloid recurrence rate will be evaluated at each visit, and the scar prevention in plastic surgery will be evaluated comparing laser treated portion and non-treated portion.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Skin type from I to VI (Fitzpatrick classification scale)
* Scar longer than 4cm for plastic surgery's patients OR scar longer than 2cm for keloid patients

Exclusion Criteria:

* Malignant tumor pathology
* Infectious or viral skin disease
* Immunosuppressive pathology and/or immunosuppressive treatment,
* Long-term corticosteroid treatment
* Pregnant woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-04 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
treatment tolerability assessed by natures, intensity and incidences of the side effects, with a special oversight of skin burn lesion | 10 days after surgery or excision

SECONDARY OUTCOMES:
improvement of scarring for plastic surgery group | 12 months after surgery
  * Vancouver Scar Scale score
  * Comparative scar assessment scale
  * Observer assessment score (POSAS)
keloid recurrence, an intralesional corticotherapy will be set up as soon as there is a recurrence. | 12 months after excision
  * Lesion size
  * Vancouver scar scale
  * Observer scar scale (POSAS)
quality of life assessment for keloid group | 12 months after excision
  * VQ-dermato
  * satisfaction questionnaire
Socio and medical economic evaluation for keloid group | 12 months after excision

CONTACTS AND LOCATIONS:
Overall Officials: Guy Magalon, MD PhD, Principal Investigator — plastic and reconstructive surgey department, APHM
Locations (1):
- Magalon, Marseille, France